CLINICAL TRIAL: NCT03069391
Title: The Interactive Physical and Cognitive Exercise System (iPACES™): A Neuro-exergame for Preventing Alzheimer's and Ameliorating Cognitive Impairment
Brief Title: The Interactive Physical and Cognitive Exercise System
Acronym: iPACES™
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Union College, New York (Other)
Collaborators: 1st Playable Productions (Other); Albany Medical College (Other); Skidmore College (Other); University of Illinois at Urbana-Champaign (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Cay Anderson-Hanley, PhD, Associate Professor, Union College, New York
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 16028; 1R41AG053120-01 (NIH)
Record Dates: First submitted 2017-02-07; First posted 2017-03-03 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Alzheimer Disease, Early Onset; MCI; Aging; Mild Cognitive Impairment; Neurocognitive Disorder; Cognitive Impairment; Cognitive Change
Keywords: exercise; exergame
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Neurocognitive Disorders; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Crossover RCT: participants are randomly assigned to start with one form of intervention and then crossover to another form of the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- physical, cognitive, then interactive (Active Comparator): physical exercise alone (PES) first, then iPACES
  Interventions: Behavioral: physical exercise alone (PES) first; Device: interactive Physical and Cognitive Exercise (iPACES™)
- cognitive, physical, then interactive (Active Comparator): cognitive exercise alone (iCE) first, then iPACES
  Interventions: Device: cognitive exercise alone (iCE) first; Device: interactive Physical and Cognitive Exercise (iPACES™)

INTERVENTIONS:
Behavioral: physical exercise alone (PES) first — following 2-week placebo for all participants, participants in this arm will then start their active intervention with a randomly assigned 2-week physical exercise-only intervention, then 2-week cognitive exercise-only intervention, then 2-week and 3 month intervals of iPACES™ (interactive physical and cognitive exercise)
  Other Names: PES
  Arms: physical, cognitive, then interactive
Device: cognitive exercise alone (iCE) first — following 2-week placebo for all participants, participants in this arm will then start their active intervention with a randomly assigned 2-week cognitive exercise-only intervention, then 2-week physical exercise-only intervention, then 2-week and 3 month intervals of iPACES™ (interactive physical and cognitive exercise)
  Other Names: iCE
  Arms: cognitive, physical, then interactive
Device: interactive Physical and Cognitive Exercise (iPACES™) — following 2-week placebo for all participants, participants in this arm will then start their active intervention with a randomly assigned 2-week cognitive exercise-only intervention, then 2-week physical exercise-only intervention, then 2-week and 3 month intervals of iPACES™ (interactive physical and cognitive exercise)
  Other Names: iPACES™

SUMMARY:
This study is intended to clarify the benefits to brain health and thinking processes that result from different forms of exercise. In particular, this study will investigate the possible benefits of physical exercise (such as pedaling an under-table stationary elliptical) or mental exercise (such as playing a videogame on a portable tablet), or combining these activities together (as in the iPACES™ exergame).

ELIGIBILITY:
Inclusion Criteria:

* co-residing older adults (e.g., spouses, partners, roommates, relatives)
* both at least 50 years of age
* normative/typical cognitive function or those with Mild Cognitive Impairment (MCI) or mild Neurocognitive Disorder (mNCD) or early Alzheimer's disease
* adequate vision and dexterity for on-screen assessments
* able to pedal an under-table elliptical
* permission of primary care provider and cardiologist (if applicable)

Exclusion Criteria:

* history of seizure
* Parkinson's disease
* significant dementia/memory loss

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-03-04 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
executive function composite score | change over time from baseline to 3 months
  comprised of scores from Stroop, Trails, and Flanker

SECONDARY OUTCOMES:
brain-derived neurotrophic factor (BDNF) | change over time from baseline to 3 months
  change in amount in saliva sample over time (pg/ml) per ELISA
Sit-Stand Test | change over time in score from baseline to 3 months
  scored performance on time and technique to move from sitting on floor to standing

CONTACTS AND LOCATIONS:
Overall Officials: Cay Anderson-Hanley, PhD, Principal Investigator — Union College
Locations (1):
- Healthy Aging & Neuropsychology Lab @ Union College, Schenectady, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wall K, Stark J, Schillaci A, Saulnier ET, McLaren E, Striegnitz K, Cohen BD, Arciero PJ, Kramer AF, Anderson-Hanley C. The Enhanced Interactive Physical and Cognitive Exercise System (iPACESTM v2.0): Pilot Clinical Trial of an In-Home iPad-Based Neuro-Exergame for Mild Cognitive Impairment (MCI). J Clin Med. 2018 Aug 30;7(9):249. doi: 10.3390/jcm7090249. PMID 30200183
- [Result] Anderson-Hanley C, Stark J, Wall KM, VanBrakle M, Michel M, Maloney M, Barcelos N, Striegnitz K, Cohen BD, Kramer AF. The interactive Physical and Cognitive Exercise System (iPACES): effects of a 3-month in-home pilot clinical trial for mild cognitive impairment and caregivers. Clin Interv Aging. 2018 Sep 4;13:1565-1577. doi: 10.2147/CIA.S160756. eCollection 2018. PMID 30233154